CLINICAL TRIAL: NCT07057115
Title: Comparison of vNOTES (Vaginal Natural Orifice Transluminal Endoscopic Surgery) Salpingectomy and Laparoscopic Salpingectomy Performed for Ectopic Pregnancy
Brief Title: Comparison of vNOTES and Laparoscopic Salpingectomy in the Surgical Treatment of Ectopic Pregnancy
Acronym: vNOTES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gopvnotesectopic
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Ectopic Pregnancy
Keywords: vNOTES; laparoscopy; salpingectomy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, parallel assignment study in which participants diagnosed with ectopic pregnancy are allocated to undergo either vNOTES salpingectomy or conventional laparoscopic salpingectomy. Randomization is performed using the envelope method. Each participant receives only one type of surgical intervention, and outcomes are compared between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vNOTES Salpingectomy Group (Experimental): Patients undergoing salpingectomy via vaginal natural orifice transluminal endoscopic surgery (vNOTES).
  Interventions: Procedure: vNOTES Salpingectomy Group.
- Laparoscopic Salpingectomy Group (Active Comparator): Patients undergoing salpingectomy via conventional laparoscopic surgery.
  Interventions: Procedure: Laparoscopic Salpingectomy

INTERVENTIONS:
Procedure: vNOTES Salpingectomy Group. — Participants will undergo salpingectomy using the vaginal natural orifice transluminal endoscopic surgery (vNOTES) technique. This minimally invasive procedure is performed transvaginally without abdominal incisions, offering potential benefits such as less postoperative pain, faster recovery, and better cosmetic outcomes.
  Arms: vNOTES Salpingectomy Group
Procedure: Laparoscopic Salpingectomy — Participants will undergo conventional laparoscopic salpingectomy, a minimally invasive surgical technique performed through small abdominal incisions using a laparoscope. This method is the current standard approach for managing ectopic pregnancies.
  Arms: Laparoscopic Salpingectomy Group

SUMMARY:
This study compares vNOTES salpingectomy and laparoscopic salpingectomy in the treatment of ectopic pregnancy, focusing on outcomes such as operative time, postoperative pain, and recovery.

DETAILED DESCRIPTION:
This study aims to compare the clinical outcomes of two surgical approaches-vaginal natural orifice transluminal endoscopic surgery (vNOTES) salpingectomy and conventional laparoscopic salpingectomy-in patients diagnosed with ectopic pregnancy. The primary objective is to evaluate and contrast parameters such as operative time, postoperative pain, complication rates, hospital stay duration, and recovery times between the two groups. The goal is to assess the feasibility, safety, and effectiveness of the vNOTES technique as an alternative minimally invasive method for the management of ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with ectopic pregnancy Without heterotopic pregnancy Women aged 18-55 years, within reproductive age Patients for whom medical treatment is not appropriate Patients requiring surgical intervention Patients without systemic diseases that may contraindicate surgery Patients who have signed and approved the informed consent form to participate in the study

Exclusion Criteria:

Ectopic pregnancy cases that can be treated with medical therapy Patients with advanced pelvic infections or pelvic anatomical abnormalities Patients with immunodeficiency or systemic diseases that contraindicate surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Function Measured by PISQ-12 at 6 Months | 6 months postoperatively
  Sexual function will be evaluated using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12), a validated instrument for assessing sexual function in women with pelvic floor disorders. Scores range from 0 to 48, with higher scores indicating better sexual function. The change in PISQ-12 scores from baseline to 6 months postoperatively will be compared between the vNOTES and laparoscopic groups.
Postoperative Pain Score (VAS) at 6 Hours After Surgery | 6 hours postoperatively
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain. The pain score at the 6th postoperative hour will be compared between the vNOTES and laparoscopic groups.

CONTACTS AND LOCATIONS:
Overall Officials: havva betül bacak, md, Principal Investigator — Gaziosmanpaşa training and research hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No